CLINICAL TRIAL: NCT00936962
Title: Evaluation of Meningococcal C Vaccine Programmes in Canadian (BC, NS, Alta.) Children During Peak Years of Risk (0-<5 Years of Age)
Brief Title: Evaluation of Meningococcal C Vaccine Programmes in Canadian Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: H07-02175
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Meningococcal Sero-type C Infection
Keywords: Meningococcal C vaccine; Meningitis study; Canadian vaccine schedule; Prevention of Meningococcal C disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 NeisVac C vaccine - 0 doses (Experimental): NeisVac C (Meningococcal C) vaccine - 0 doses
  Interventions: Biological: NeisVac C vaccine (12mth)
- Group 2 NeiscVac C - 2 doses (Experimental): 2 priming doses of NeisVac C vaccine at 2 and 4 mths of age
  Interventions: Biological: NeisVac C vaccine (12mth)
- Group 3 NeiscVac C - 1 dose (Experimental): 1 priming dose of NeisVac C vaccine at 2 mths of age
  Interventions: Biological: NeisVac C vaccine (12mth)

INTERVENTIONS:
Biological: NeisVac C vaccine (12mth) — NeisVac C Meningococcal C Conjugate vaccine given IM 0.5mL in the deltoid muscle at 12 mths of age
  Other Names: NeisVac C vaccine (Baxter); Meningococcal C congugate vaccine

SUMMARY:
The purpose of the study is to see which of the three current provincial Meningococcal C Conjugate vaccine schedules in Canada provide the longest lasting protection against Meningococcal C disease and to see if a booster vaccination is needed.

DETAILED DESCRIPTION:
In 2002-2005, Canada introduced universal MenC programmes consisting of 1,2 or 3 infant doses. Most are one (12 mth) dose. High rates of serogroupC disease in 2000 and 2001 prompted some provinces to launch universal MenC vaccination programmes in 2002. The goal was to provide protection in infancy and early childhood (the time of most risk) with the hope that the protection would extend throughout adolescence (the second highest risk). It is unclear if early multi-dosing or 1 dose programmes would offer better protection (lack of data). Each province in Canada has chosen different Meningococcal C Conjugate vaccine provision schedules for the primary vaccinations.

This study will look at short term protection after the differing provincial series of vaccinations has been given and compare those who do not get primary vaccination under 1 year of age (NS) with two schedules of primary immunization (BC at 2 and 4 mths and Alberta at 2 months). A blood sample will be collected at 12-13 mths for this comparison. A booster vaccination of the current provincial Men C vaccine will be provided at 12 months. Another blood sample will be collected 1 mth later to look at the difference in responses between the groups (different provincial primary vaccination schedule). 2 years and 4 years later (at age 3 and age 5), another blood sample will be collected to look at the difference in long term protection of the groups where the primary schedule was different.

ELIGIBILITY:
Inclusion Criteria:

* 12-13 mths of age
* over 34 weeks gestation
* healthy children
* having had all vaccinations of Meningococcal C vaccine per the recommended schedule for their respective province within a month of the recommended age - documented.
* Communication in English

Exclusion Criteria:

* No contraindication to receiving 12 mth dose of MenC vaccine
* No other MenC vaccine or MenC disease

Ages: 12 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 452 (Actual)
Dates: Start 2009-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the longest lasting protection against Meningococcal C disease and to see if a booster vaccination is needed. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bettinger, Ph.D, Principal Investigator — University of British Columbia; David Scheifele, Ph.D, Study Director — University of British Columbia; Scott Halperin, Ph.D, Study Director — Dalhousie University, Halifax; James Kellner, Ph.D, Study Director — University of Calgary
Locations (3):
- Canada (3):
  - Alberta Health Services (Alberta Children's Hospital), Calgary, Alberta
  - Vaccine Evaluation Center (University of BC at Children's Hospital), Vancouver, British Columbia
  - Canadian Centre for Vaccinology (Dalhousie/IWK,), Halifax, Nova Scotia

REFERENCES:
- [Derived] Bettinger JA, Scheifele DW, Halperin SA, Kellner JD, Vanderkooi OG, Schryvers A, De Serres G, Alcantara J. Evaluation of meningococcal serogroup C conjugate vaccine programs in Canadian children: interim analysis. Vaccine. 2012 Jun 8;30(27):4023-7. doi: 10.1016/j.vaccine.2012.04.034. Epub 2012 Apr 23. PMID 22537988
- See also: click here for information on the trial — http://www.vec.med.ubc.ca
- See also: Click here for interim analysis publication — http://www.ncbi.nlm.nih.gov/pubmed/22537988